CLINICAL TRIAL: NCT04987931
Title: Real-World Patient Characteristics, Treatment Patterns, and Clinical Outcomes Among Talazoparib-Treated Patients With HER2-Negative, Locally Advanced or Metastatic Breast Cancer and Germline BRCA1/2 Mutations: US Chart Review
Brief Title: Real-World Outcomes of US Talazoparib-Treated Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C3441053
Record Dates: First submitted 2021-07-14; First posted 2021-08-03 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Talazoparib; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary population: Talazoparib-treated patients with HER2- ABC with gBRCA1/2m: HER2-negative ABC patients with gBRCA1/2 mutations treated with talazoparib monotherapy initiated on or after October 16, 2018 and ≥18 years of age at initiation of talazoparib.
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — This retrospective chart review study focuses on patients with HER2- ABC with gBRCA1/2m initiating talazoparib on or after October 16, 2018 and ≥18 years of age at initiation of talazoparib.
  Other Names: TALZENNA®

SUMMARY:
This study is a retrospective, multi-site, patient-level medical chart review of US adult patients with locally advanced or metastatic breast cancer (ABC) who initiated talazoparib on or after October 16, 2018 and were managed by participating providers from Cardinal Health's Oncology Provider Extended Network (OPEN).

This study will describe patient characteristics, treatment patterns, and clinical outcomes of talazoparib-treated patients in real-world practice setting in US.

The primary population for this study includes:

-HER2-negative ABC patients with germline BRCA1/2 (gBRCA1/2) mutations treated with talazoparib monotherapy initiated on or after October 16, 2018 and ≥18 years of age at initiation of talazoparib.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with HER2-negative ABC
* gBRCA1/2 mutation(s)
* Treatment with talazoparib monotherapy initiated on or after October 16, 2018

  -≥18 years of age at initiation of talazoparib
* A minimum of 6 months follow-up time after initiation of talazoparib unless the patient died within this follow-up period

Exclusion Criteria:

* Participation in any BC clinical trial after initiation of talazoparib
* Treatment with a PARP inhibitor as neoadjuvant/adjuvant therapy
* gBRCA1/2 or HER2 status unknown
* Diagnosis of any other malignancy, except carcinoma in situ or nonmelanoma skin cancer, within the 5 years prior to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The primary population for this study includes:
  -HER2-negative ABC patients with germline BRCA1/2 (gBRCA1/2) mutations treated with talazoparib monotherapy initiated on or after October 16, 2018 and ≥18 years of age at initiation of talazoparib.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3441053

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with human epidermal growth factor receptor 2 (HER2)-negative advanced breast cancer (ABC) germline breast cancer susceptibility gene 1 or gene 2 mutations (gBRCA 1/2m), who initiated treatment with talazoparib on or after 16-October-2018 till 11-Oct-2021 (approximately 36 months) and were greater than or equal to (>=) 18 years of age during treatment initiation were observed retrospectively in this study.
Pre-assignment Details: Data from eligible participants were retrieved and observed in this retrospective chart review study from 20-August-2021 to 11-October-2021 (approximately 1.7 months of this study). Participants were managed by physicians from Cardinal Health's Oncology Provider Extended Network (OPEN).
Groups:
- Talazoparib: Eligible participants who initiated treatment with talazoparib for HER2- ABC gBRCA 1/2m on or after 16-Oct-2018 were included.
Period: Overall Study
Arm/Group | Talazoparib
Started | 84
Completed | 84
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants with HER2- ABC gBRCA 1/2m who initiated talazoparib on or after 16-October-2018 and were >=18 years of age at initiation of talazoparib.
Arm/Group | Talazoparib
Number analyzed (Participants) | 84
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 14
  White | 60
  More than one race | 0
  Unknown or Not Reported | 5
Number of Participants According to Molecular Sub-Types of HER2- ABC gBRCA 1/2m [Count of Participants; unit: Participants] — Number of participants with HER2-ABC gBRCA 1/2m were classified according to their molecular sub-types as HR+HER2-ABC gBRCA 1/2m and triple negative breast cancer (TNBC) gBRCA 1/2m.
  Participants
    HR+ HER2- ABC gBRCA1/2 m | 30
    TNBC gBRCA 1/2m | 54
Line of ABC Therapy in Which Talazoparib was Initiated [Count of Participants; unit: Participants] — The number of participants were classified according to line of ABC therapy in which talazoparib was initiated.
  Participants
    First | 12
    Second | 34
    Third | 29
    Fourth | 9

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure (TTF) for Talazoparib
Description: TTF was defined as the time from initiation of talazoparib to discontinuation for any reason, which included disease progression, treatment toxicity, and death. Index date was defined as the date of initiation of talazoparib on or after 16-October-2018. Median was analyzed using the Kaplan-Meier method.
Time Frame: Index date up to talazoparib discontinuation, from 16-October-2018 maximum up to 11-October-2021 (approximately 36 months); data retrieved and studied from 20-August-2021 to 11-October-2021 (approximately 1.7 months of this study)
Population: Analysis population included all eligible participants with HER2- ABC gBRCA 1/2m who initiated talazoparib on or after 16-October-2018 and were >=18 years of age at initiation of talazoparib. Here ''Overall Number of Participants Analyzed'' signifies number of participants with TTF event.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 52
Months | 8.5 [8.0 to 9.7]

2. Secondary Outcome: Real-World Progression Free Survival (rwPFS) From Initiation of Talazoparib
Description: rwPFS was defined as the time from initiation of talazoparib to charted disease progression based on radiographic imaging or death from any cause, whichever occurred first. Index date was defined as the date of initiation of talazoparib on or after 16-October-2018. Since information was retrieved from participants' charts, there was no specific criteria for progression. It was determined on physician judgement. Median was analyzed using the Kaplan-Meier method.
Time Frame: Index date up to charted disease progression, from 16-October-2018 maximum up to 11-October-2021 (approximately 36 months); data retrieved and studied from 20-August-2021 to 11-October-2021 (approximately 1.7 months of this study)
Population: Analysis population included all eligible participants with HER2- ABC gBRCA 1/2m who initiated talazoparib on or after 16-October-2018 and were >=18 years of age at initiation of talazoparib. Here ''Overall Number of Participants Analyzed'' signifies number of participants with rwPFS event.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 52
Months | 8.7 [8.0 to 9.9]

3. Secondary Outcome: Time From Initiation of Talazoparib to Initiation of Subsequent Chemotherapy
Description: The time taken for initiating subsequent chemotherapy after initiation of talazoparib was reported in this outcome measure. Index date was defined as the date of initiation of talazoparib on or after 16-October-2018. Median was analyzed using the Kaplan-Meier method.
Time Frame: Index date up to initiation of subsequent chemotherapy, from 16-October-2018 maximum up to 11-October-2021 (approximately 36 months); data retrieved and studied from 20-August-2021 to 11-October-2021 (approximately 1.7 months of this study)
Population: Analysis population included all eligible participants with HER2- ABC gBRCA 1/2m who initiated talazoparib on or after 16-October-2018 and were >=18 years of age at initiation of talazoparib. Here ''Overall Number of Participants Analyzed'' signifies number of participants with chemotherapy after talazoparib initiation.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Talazoparib
Number analyzed (Participants) | 21
Months | 12.2 [10.5 to 20.1]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: index date up to death due to any cause, from 16-October-2018 maximum up to 11-October-2021 (approximately 36 months); data retrieved and studied from 20-August-2021 to 11-October-2021 (approximately 1.7 months of this study); since adverse events (AEs) were not collected hence time frame for AEs not applicable
Description: AEs were not collected during the retrospective chart review of this study.
Arm/Group | Talazoparib
All-Cause Mortality (participants affected / at risk) | 38/84
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT04987931/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-10): https://cdn.clinicaltrials.gov/large-docs/31/NCT04987931/SAP_001.pdf